CLINICAL TRIAL: NCT04385134
Title: Establishment and Application of the National Surveillance Network for Enterovirus During the Perinatal Period
Brief Title: Enterovirus Surveillance During the Perinatal Period
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bayi Children's Hospital Affiliated to PLA Army General Hospital, China (Other)
Responsible Party: Sponsor
Organization: Seventh Medical Center of PLA General Hospital (Other)
Other Study IDs: Bayichildren's-02
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Enterovirus Infection During Perinatal Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- General parturient: Observe the enterovirus infection in general parturients and their neonates.
  Interventions: Other: No intervention
- Puerpera with fever: Observe the enterovirus infection in puerpera with fever and their neonates.
  Interventions: Other: No intervention
- Febrile newborns: Observe the enterovirus infection in neonates
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Neonates could be infected by non-polio enterovirus easily. Some of the neonates may develop fatal complications within one week. The objective of this study were as following: 1.To understand the composition and epidemiological characteristics of enterovirus infection in pregnant women in some areas of China; 2.To understand the transmission from mother to their neonates; 3.To understand the pathogenic spectrum composition, epidemiological characteristics and clinical characteristics of enterovirus infection in neonates; 4.To understand the genetic variation and changes of enteroviruses; 5.To establish a quality management system for maternal and neonatal enterovirus laboratory testing and monitoring.

ELIGIBILITY:
Inclusion Criteria:

* 1. General parturient: on the first day of the third week of each month, all parturients and their newborns admitted to the hospital (day shift 8:00-18:00) within that day; 2. Puerpera with fever: all puerperas with fever (body temperature >=37.5 degree C) and their newborns were included in summer and autumn (from May); 3. Febrile newborns: those included in summer and autumn (from May) with the following clinical characteristics: fever >=37.5 degree C, lasting for more than one day. And sign the informed consent form with the consent of the guardian.

Exclusion Criteria:

* 1. Pregnant women with urinary tract infection, chorioamnionitis and bacterial infection; 2. Puerpera with fever due to urinary tract infection, chorioamnionitis and bacterial infection; 3. Newborns infected with other pathogens.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Three population would be studied. 1. General parturient; 2. Puerpera with fever; 3, Febrile newborns.
Sampling Method: Probability Sample
Enrollment: 6500 (Estimated)
Dates: Start 2020-05-20 (Estimated); Primary Completion 2021-05-20 (Estimated); Study Completion 2022-12-25 (Estimated)

PRIMARY OUTCOMES:
Detection of enterovirus | 42 days
  Detection of the rate of enterovirus infection and identify the genotype of enterovirus.

SECONDARY OUTCOMES:
Detection of antibodies of enterovirus | 42 days
  Detection of IgG antibodies of enterovirus

CONTACTS AND LOCATIONS:
Locations (1):
- Bayi Children's Hospital, Seventh Medical Center, PLA general hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No